CLINICAL TRIAL: NCT05423561
Title: Sclerotic Bone Formation (Corticalisation) on the Intramedullar Nail Tip in Hypertrophic Non-union Developing After Femoral Transverse Diaphyseal Fractures
Brief Title: Corticalisation After Femoral Nail Dynamization in Hypertrophic Non-unions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Ali Çağrı Tekin, Associated Professor, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-48670771-514.99; 67 (Registry Identifier: Desicion number)
Record Dates: First submitted 2022-06-09; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Pseudoarthrosis of Bone; Implant Breakage
Keywords: hypertrophic pseudarthrosis; dynamization; corticalisation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- hypertrophic non-union developing after femoral transverse diaphyseal fractures (Other)
  Interventions: Procedure: exchange nailing with larger, thicker nail crossing corticalization

INTERVENTIONS:
Procedure: exchange nailing with larger, thicker nail crossing corticalization — exchange nailing with larger, thicker nail crossing corticalization

SUMMARY:
In 12 patients with corticalization and hypertrophic pseudarthrosis were present after dynamization, the old nail was removed and nail exchange was performed with a longer and larger diameter nail to pass the region formed in the cortex approximately 2-3cm inferior from the old nail.

DETAILED DESCRIPTION:
Corticalization is cortex-like sclerosis in the distal of the nail and it may indicate the early sign of dynamization treatment failure in hypertrophic nonunion after femoral transverse diaphyseal fractures. When corticalization is seen during follow-up after dynamization is performed because of non-union of a femoral transverse fracture, nail exchange should be performed without further delay. More rigid fixation should be applied with a longer and thicker nail crossing the area of corticalization.

ELIGIBILITY:
Inclusion Criteria:

* Subtrochanteric fractures
* Nonunion with Pain

Exclusion Criteria:

* Infection
* Pathological Fracture (Tumor)

Ages: 28 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Provide Bone Union | 6 months
  Achievement of bone union with detecting callus formation on radiography after passing the region of corticalisation with a longer and thicker nail
Relieving pain in the nonunion area | 6 weeks
  Detection of reduction of pain scores in the nonunion area and enabling patients to load on the extremity in the early period postoperatively

IPD SHARING:
Plan to Share IPD: No